CLINICAL TRIAL: NCT07371754
Title: Shear Wave Elastography of Intercostal Muscles for the Non-invasive Assessment of the Work of BreathinG
Acronym: SWING
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A01528-41
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COPD; Healthy Adult
Keywords: Shear wave elastography; Intercostal muscles; work of breathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy adults: Participant without respiratory, muscle or thoracic abnormalities
  Interventions: Diagnostic Test: Intercostal muscle shear wave elastography (SWE) during standardized inspiratory loading
- COPD group: Patients with COPD
  Interventions: Diagnostic Test: Intercostal muscle shear wave elastography (SWE) during standardized inspiratory loading

INTERVENTIONS:
Diagnostic Test: Intercostal muscle shear wave elastography (SWE) during standardized inspiratory loading — Ultrasound shear wave elastography (SWE) is performed to quantify intercostal muscle stiffness at rest and during standardized inspiratory loading/controlled breathing. SWE acquisitions are synchronized with physiological reference recordings (e.g., esophageal pressure and/or diaphragm EMG when available) to estimate and track respiratory effort/work noninvasively.
  Other Names: Ultrasound shear wave elastography of intercostal muscles

SUMMARY:
Quantifying respiratory effort is a key step in physiological and clinical research on exercise tolerance, mechanisms of fatigability, and ventilatory impairment. To date, reliable assessment relies on an invasive method: esophageal pressure (Pes) measurement using a balloon catheter inserted into the esophagus. Although Pes provides an indirect estimate of pleural and intrathoracic pressure, it is uncomfortable for patients, requires dedicated equipment, and may limit study participation.

In critically ill patients, a noninvasive approach to quantify respiratory effort would have major clinical and scientific value. In acute respiratory distress, accurately tracking the intensity and evolution of respiratory effort could support earlier therapeutic decision-making.

Shear Wave Elastography (SWE) is an ultrasound technology enabling very high acquisition rates and estimating tissue stiffness from shear-wave propagation induced by an acoustic impulse. Because muscle stiffness is strongly related to force produced during contraction, we hypothesize that intercostal muscle stiffness measured by SWE correlates with respiratory work and increases with rising inspiratory load.

ELIGIBILITY:
Inclusion Criteria:

Adult patient with chronic obstructive pulmonary disease (COPD), stage 3-4.

Healthy adult volunteer.

Exclusion Criteria:

Refusal to participate or withdrawal of consent.

Age < 18 years.

BMI > 35 kg/m².

Pregnancy or breastfeeding.

Inability to understand instructions or cooperate (cognitive impairment, language barrier).

Neurological condition affecting breathing (e.g., recent stroke, ALS, myopathy).

Thoracic condition limiting access to the intercostal muscles (e.g., major chest wall deformity, surgical scar).

Recent thoracic or abdominal surgery (< 3 months).

Known esophageal disease (stricture, achalasia, severe esophagitis, diverticulum, history of perforation).

ENT or tracheal abnormality preventing probe insertion (e.g., tumor, malformation, tracheostomy).

Swallowing disorders or risk of aspiration.

Recent exacerbation (< 6 weeks).

Oxygen therapy > 2 L/min during exertion.

Hemodynamic instability.

Not affiliated with a social security scheme.

Legally protected persons (as defined by law).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) will be enrolled in two cohorts: (1) healthy adult volunteers and (2) adult patients with chronic obstructive pulmonary disease (COPD), stage 3-4. A total of 20 participants will be recruited (10 COPD patients and 10 healthy volunteers). Each participant will complete a single study visit (~45 minutes) involving standardized breathing/inspiratory loading while intercostal muscle ultrasound shear wave elastography is recorded, with concurrent physiological reference measurements to quantify respiratory effort.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between intercostal muscle stiffness (SWE) and respiratory effort (esophageal pressure-time product) | During a single study visit (≈45 minutes), at rest and at each standardized inspiratory load level
  Intercostal muscle stiffness (kPa) measured by shear wave elastography is correlated with respiratory effort quantified by the esophageal pressure-time product (PTPes; cmH2O·s/min) across the standardized inspiratory loading protocol (within each cohort).

SECONDARY OUTCOMES:
Within-subject change in intercostal muscle stiffness (SWE) across inspiratory load levels | Single study visit: during the inspiratory loading protocol (no resistance, then 25%, 50%, and 75% of maximal inspiratory pressure [PiMax])
  Intercostal muscle stiffness (kPa) measured by shear wave elastography (SWE) will be assessed within participants across the different inspiratory load levels.

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request. Requests will be reviewed on a case-by-case basis and, if approved, de-identified data and relevant documentation (e.g., protocol and data dictionary) will be shared under an appropriate data use agreement.